CLINICAL TRIAL: NCT03063099
Title: A Pilot Study of ReNu™ Hip Injection: Monitoring the Response of Hip Function and Pain in Patient With Osteoarthritis
Brief Title: ReNu™ Injection to Treat Hip Osteoarthritis Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NuTech Medical, Inc (Industry)
Collaborators: Organogenesis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD2016-01-01
Record Dates: First submitted 2017-02-21; First posted 2017-02-24 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ReNu™ Injection (Experimental): ReNu™ is an allograft tissue composed of particularized amniotic membrane and cell from the amniotic fluid.
  Interventions: Other: ReNu™ Injection

INTERVENTIONS:
Other: ReNu™ Injection — Injection into the hip for the treatment of Osteoarthritis.

SUMMARY:
A pilot study to evaluate changes in hip function and pain in patients with osteoarthritis receiving the ReNu™ Hip Injection.

DETAILED DESCRIPTION:
This is a prospective, non-randomized pilot study evaluating the efficacy of ReNu™ hip injection on patients with moderate osteoarthritis. The effects will be measured primarily through patient-reported outcomes questionnaires after a single injection. Patients will be followed up to 12 months to evaluate improvements using common pain and function subscales.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate hip osteoarthritis determined by a combination of clinical and radiographic findings
* Radiographic findings consistent with osteoarthritis as documented by Tonnis radiographic classification (Grade 1 or 2)
* Grade 1 Tonnis changes are defined as mild and include increased sclerosis, slight narrowing of the joint space, no or slight loss of head sphericity
* Grade 2 Tonnis changes are defined as moderate and include small cysts, moderate narrowing of the joint space, moderate loss of head sphericity
* Patients with bilateral grade 1or 2 Tonnis hip osteoarthritis who have bilateral symptoms may have their more symptomatic hip injected. If equivalent symptoms are reported by the patient, then the patient will choose which hip is to be injected. The other Hip can be treated with all standard local interventions that will not have a prolonged systemic effect that could affect the study hip (for example steroid injection, cold therapy, soft braces).
* Between the Ages 18 to 70 with minimum activity level of 2 on the Tegner scale.
* BMI less than 40
* Female patients must be actively practicing a contraception method, abstinence, be surgically sterilized, or be postmenopausal

Exclusion Criteria:

* Pain medication (including NSAIDs) less than 15 days before injection (may take acetaminophen)
* Receiving pain medication other than acetaminophen for conditions unrelated to osteoarthritis of the index hip
* Regular use of anticoagulants, such as Coumadin, dabigatran or rivaroxaban; use of antiplatelet medications are not a reason for exclusion
* History of substance abuse.
* Failure to agree NOT to take additional hip symptom modifying drugs, other than acetaminophen, during the course of the study without reporting to the study team
* Pregnancy or desire to become pregnant during study duration
* Corticosteroid injection into the index hip within 6 months
* Viscosupplement injection into the index hip within 6 months
* Previous open or arthroscopic hip surgery of the involved index hip within the previous 6 months
* Open or arthroscopic surgery of the contralateral hip within the last 6 months
* Worker compensation
* Acute index hip injury (injury within 3 months)
* History of Diabetes mellitus
* History of solid organ or hematologic transplantation
* History of rheumatoid arthritis or other autoimmune disorder
* Diagnosis of a non-basal cell malignancy within the preceding 5 years
* Infection requiring antibiotic treatment within the preceding 3 months
* Current therapy with any immunosuppressive medication, including corticosteroids at a dose > 5 mg per day

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
IHOT12 - International Hip Outcome Tool 12 | 3 & 6 months
  Change from Baseline
Visual Analog Scale (VAS) Pain Scale | 3 & 6 months
  Change from Baseline

SECONDARY OUTCOMES:
Modified Harris Hip Score | 3, 6 & 12 months
  Change from Baseline
SF12 Score | 3, 6 & 12 months
  Generic measure of patient's health status change from baseline
Single Assessment Numerical Evaluation (SANE) | 3, 6 & 12 months
  Measurement tool used to record patient's self-reported change in function from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Katie Mowry, PhD, Study Director — Organogenesis
Locations (2):
- United States (2):
  - Stanford Medicine Orthopaedic Surgery, Redwood City, California
  - Rush University Medical Center, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No